CLINICAL TRIAL: NCT01730677
Title: Randomized Phase II Study of Lapatinib Plus Vinorelbine Versus Vinorelbine in Patients With HER2 Positive Metastatic Breast Cancer Progressed After Lapatinib and Trastuzumab Treatment
Brief Title: Lapatinib+Vinorelbine vs Vinorelbine HER2 Positive Metastatic Breast Cancer Progressed After Lapatinib/Trastuzumab
Acronym: LV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Asan Medical Center (Other); Chung-Ang University (Other); Korea University Anam Hospital (Other); Samsung Medical Center (Other); Seoul National University Hospital (Other); Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jungsil Ro, Chief, Center for Clinical Trials, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-11-583
Record Dates: First submitted 2012-07-15; First posted 2012-11-21 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Metastatic Breast Cancer
Keywords: Lapatinib; Vinorelbine
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lapatinib+Vinorelbine (Experimental): lapatinib 1000mg, once daily vinorelbine 20mg/m2, D1 and D8, every 3 weeks
  Interventions: Drug: Lapatinib; Drug: Vinorelbine
- Vinorelbine (No Intervention): vinorelbine 30mg/m2, D1 and D8, every 3 weeks

INTERVENTIONS:
Drug: Lapatinib — lapatinib 1000mg, once daily
  Other Names: LV arm
  Arms: Lapatinib+Vinorelbine
Drug: Vinorelbine — Vinorelbine 20mg/m2, D1 and D8, every 3 weeks
  Other Names: LV arm
  Arms: Lapatinib+Vinorelbine

SUMMARY:
The investigators address the clinical efficacy of continuing lapatinib treatment combined with vinorelbine after the progression of both trastuzumab and lapatinib treatment compared with vinorelbine alone in HER2 positive metastatic breast cancer patients.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, open label, phase II study. Patients will be randomized to either lapatinib plus vinorelbine (LV) arm or vinorelbine alone (V) arm, if they are satisfied by inclusion and exclusion criteria. The stratification factors are followings: 1) visceral metastasis vs. others, 2) previous response to lapatinib treatment, complete response(CR)+partial response(PR) vs. stable disease(SD)≥ 12wks.

Patients in LV arm will receive daily lapatinib 1,000mg with vinorelbine 20mg/m2 day1 and day 8. Patients in V arm will receive vinorelbine 30mg/m2 day 1 and day 8. Treatment repeats every 21 days unless there is any evidence of disease progression or unacceptable toxicity or noncompliance by patient with protocol requirements. Response will be documented by physical examination, chest or abdomen CT prior to treatment as a baseline, and every 2 cycles (window period ± 1 week) after a start of treatment and at 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed stage IV or recurrent breast cancer
* Documented HER2 status and positive for HER2 in tumor cells by immunohistochemistry (3+) or FISH (The results of SISH or CISH are also allowed)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Age ≥ 20 years
* Measurable or evaluable disease according to the Response Evaluation Criteria in Solid Tumors version 1.1
* Patients who were treated with anthracycline based regimens in the adjuvant/neoadjuvant or metastatic setting.
* Patients who experienced disease progression after the treatment with lapatinib containing regimens whose response were more than stable disease (including CR, PR, SD≥ 12 weeks) during treatment. There is no limitation on the time interval between the stop of lapatinib treatment and the study enrollment.
* Patients must have received 2 or 3 lines of prior anti-HER2 therapy in metastatic setting as follows regardless of the order
* In case with trastuzumab: monotherapy or combined with taxane or combined with AI
* In case with lapatinib: monotherapy or combined with capecitabine or combined with AI
* Patients who received T-DM1 or pertuzumab with trastuzumab previously are allowed in this study
* Patients who received neratinib, mTOR inhibitor, PI3K/AKT inhibitor, or BIBW2992 are not eligible
* Patients who experienced a disease recurrence during receiving adjuvant trastuzumab or within 6 months after the completion of adjuvant trastuzumab treatment are allowed even when patients did not receive trastuzumab in the metastatic setting.
* Patients who experienced a disease recurrence during receiving adjuvant lapatinib or within 6 months after the completion of adjuvant lapatinib treatment are allowed as long as they meet criteria of CR, PR or SD ≥ 12 weeks by lapatinib/capecitabine treatment for metastatic disease.
* Central nervous system metastasis is permitted if asymptomatic or controlled with minimal steroid requirement and is documented to be non-progressing at study entry.
* Negative urine pregnancy test within 7 days prior to registration in premenopausal patients
* Baseline LVEF ≥50% measured by echocardiogram or multiple gated acquisition scan (MUGA) scan
* Adequate hematopoietic function: Absolute granulocyte count ≥1,500/mm3, platelet≥100,000/mm3, hemoglobin≥9g/mm3
* Adequate hepatic function: total bilirubin ≤1.5mg/dL, AST/ALT≤2 x upper normal limit (UNL), alkaline phosphatase ≤2.5 x UNL, in case with bone metastases alkaline phosphatase ≤5 x UNL
* Adequate renal function: Serum creatinine ≤1.5mg/dL
* Ability to understand and comply with protocol during study period
* Patients should sign a written informed consent before study entry

Exclusion Criteria:

* Pregnant or lactating women or women of childbearing potential, including women whose last menstrual period was ,12 months ago (unless surgically sterile) who are unable or unwilling to use adequate contraceptive measures during the study treatment period.
* Patients who received vinorelbine treatment in metastatic setting.
* Patients who received more than 3 lines of prior anti-HER2 therapy in metastatic setting
* Patients who have history of cancer other than in situ uterine cervix cancer or nonmelanotic skin cancer
* Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled GI disease (e.g., Crohn's disease, ulcerative colitis)
* current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Concurrent disease or serious medical disorder,
* Serious cardiac illness :

History of documented congestive heart failure (CHF) or systolic dysfunction (LVEF <50%) High-risk uncontrolled arrhythmias (ventricular tachycardia, high-grade atrioventricular (AV)-block,supraventricular arrhythmias, prolonged corrected QT (QTc) which are not adequately rate-controlled) Angina pectoris requiring antianginal medication Clinically significant valvular heart disease Evidence of transmural infarction on ECG Poorly controlled hypertension (e.g. systolic >180mm Hg or diastolic >100mm Hg)

- known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to any of the study agents or their excipients.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival rate at 18 weeks | The time point of 18 weeks from the initiation of study treatment.
  The PFS rate at 18 weeks will be calculated as the ratio of patients on the study to Intent to treat (ITT) population at the time point of 18 weeks from the initiation of study treatment. The ITT population will consist of all patients who are randomized.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From date of randomization until the date of first documented progression, withdrawal from the study, or date of death from any cause, whichever came first, assessed up to 36 months
  The secondary objective of this study is to estimate the PFS and OS in both arms and median PFS and OS will be estimated by Kaplan-Meier estimates and compared by log-rank test. Response rate will be calculated as the proportion of patients with a complete or partial tumor response among ITT population. Chi-square test will be used to PFS rate and compare response rates between the two arms (categorical variables).
Overall survival (OS) | From date of randomization until the date of death from any cause, assessed up to 36 months
  The secondary objective of this study is to estimate the OS in both arms will be estimated by Kaplan-Meier estimates and compared by log-rank test.
toxicity | From date of randomization until the date of first documented progression, withdrawal from the study, or date of death from any cause, whichever came first, assessed up to 36 months
  All toxicities during treatment will be recorded according to NCI-common toxicity criteria for adverse effects version 4.0.
response rate | From date of randomization until the date of first documented progression, withdrawal from the study, or date of death from any cause, whichever came first, assessed up to 36 months
  Objective response mean complete response and partial response according to Response evaluation criteria in solid tumors v 1.1 and response will be assessed every 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jungsil Ro, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Sim SH, Park IH, Jung KH, Kim SB, Ahn JH, Lee KH, Im SA, Im YH, Park YH, Sohn J, Kim YJ, Lee S, Kim HJ, Chae YS, Park KH, Nam BH, Lee KS, Ro J. Randomised Phase 2 study of lapatinib and vinorelbine vs vinorelbine in patients with HER2 + metastatic breast cancer after lapatinib and trastuzumab treatment (KCSG BR11-16). Br J Cancer. 2019 Dec;121(12):985-990. doi: 10.1038/s41416-019-0618-z. Epub 2019 Nov 6. PMID 31690831